CLINICAL TRIAL: NCT03275064
Title: A Two-part, Randomized, Placebo-controlled, Patient and Investigator Blinded, Study Investigating the Safety, Tolerability and Preliminary Efficacy of Intra-articular LNA043 Injections in Regenerating the Articular Cartilage of the Knee in Patients With Articular Cartilage Lesions (Part A) and in Patients With Knee Osteoarthritis (Part B).
Brief Title: Study of Safety, Tolerability, Preliminary Efficacy of Intra-articular LNA043 Injections in Patients With Articular Cartilage Lesions and Knee Osteoarthritis.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CLNA043X2202; 2016-004052-30 (EudraCT Number); CTI-194705 (Other: Japic CTI)
Record Dates: First submitted 2017-08-29; First posted 2017-09-07 (Actual); Results first posted 2024-02-14 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Osteoarthritis
Keywords: Articular cartilage; partial thickness cartilage lesion; knee cartilage; regeneration; osteoarthritis; adult
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Intervention Model Description: A total of 142 participants were randomized, but only 141 received treatment. One participant in Part B was discontinued due to poor veins that were not adequate for blood samples.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- LNA043 40 mg Part B (Experimental): LNA043 40 mg Part B
  Interventions: Biological: LNA043
- LNA043 20 mg Part B (Experimental): LNA043 20 mg Part B
  Interventions: Biological: LNA043
- LNA043 20 mg Part A (Experimental): LNA043 20 mg Part A
  Interventions: Biological: LNA043
- Placebo Part A (Placebo Comparator): Placebo Part A
  Interventions: Other: Placebo
- Placebo Part B (Placebo Comparator): Placebo Part B
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: LNA043 — LNA043 intra-articular injection
  Arms: LNA043 20 mg Part A; LNA043 20 mg Part B; LNA043 40 mg Part B
Other: Placebo — Placebo intra-articular injection
  Arms: Placebo Part A; Placebo Part B

SUMMARY:
The purpose of this two-part study is to assess the efficacy, safety and tolerability of multiple intra-articular (i.a.) injections of LNA043, in regenerating the articular surface in patients with cartilage lesions of the knee (Part A) and knee osteoarthritis (Part B).

DETAILED DESCRIPTION:
There was a 30 day screening period for both Part A and Part B. In Part A, participants were randomized to 3:1 ratio and received an injection of LNA043 (20 mg in 3 ml) or matching placebo (3 ml) on Days 1, 8,15 and 22 and were monitored in clinic for 3 hours after each injection followed by telephone calls 48 hours after injection. Participants returned to the clinic on Days 50, 106, 190 and 365 for follow up visits. MRIs, safety assessments and pharmacokinetics were assessed at selected clinic visits.

In Part B, this study aimed at further evaluating the cartilage anabolic activity of LNA043 in a more severe knee OA population, and to explore the safety and efficacy of a higher dose.

In Part B, participants were randomized to LNA043 20 mg, LNA043 40 mg or matching placebo according in a 1:1:1 ratio. Injections were given in clinic on Days 1, 29, 57 and 85 and participants were monitored in clinic for 3 hours after each injection followed by telephone calls 48 hours after injection. Participants returned to the clinic on Days 113,197 and 365 (end of study) for follow up visits. MRIs, safety assessments and pharmacokinetics were assessed at selected clinic visits.

ELIGIBILITY:
Inclusion criteria Part A

* Patient was ≥18 and ≤55 years old at time of screening.
* Patient had a body mass index (BMI) <30 kg/m2 at screening,
* Patient had a symptomatic, single, articular cartilage defect of one knee, grade II or IIIA according to the ICRS classification, localized to either the femoral condyles/femoral trochlea or to the patella, based on MRI or arthroscopy performed within 9 months before screening visit and confirmed by screening 3T MRI.
* Patient had an onset of pain and impairment of function between two (2) months and two (2) years before screening.
* Patient had a grade 2 or 3 OA of the knee with Joint Space Width (JSW) 2-4 mm evaluated with X-Ray at screening

Inclusion criteria Part B

* Patient was ≥18 and ≤75 years old at time of screening.
* Patient had a body mass index (BMI) ≤ 35 kg/m2 at screening
* Diagnosis of femorotibial osteoarthritis (OA) in the target knee by standard American College of Rheumatology (ACR) criteria at study start (clinical AND radiographic criteria)
* Patient must have had symptomatic disease predominantly in one (the index) knee, with minimal or no symptoms in the contralateral knee. Symptomatic disease is defined as having pain in the knee more than 50% of the days during the last 3 months from screening.
* Patient had a K&L grade 2 or 3 OA of the knee with JSW 2.00-4.00 mm (X=0.225) fixed position evaluated with X-Ray by the Central Reader at screening.

Exclusion criteria Part A & B

* Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless they are using highly effective methods of contraception during dosing and for 15 days after stopping of investigational drug.
* Patient had surgical treatment of the target knee using mosaicplasty, microfracture, meniscectomy >50% (Note: prior diagnostic arthroscopy with debridement and lavage, <50% meniscectomy, lateral release, patellar realignment, medial patellofemoral ligament reconstruction are acceptable if performed at least 2 months prior to screening; anteriorcruciate ligament reconstrucion is acceptable if performed 12 months prior to screening, or less if restoration of joint function is evident, and agreed by the sponsor).
* Patient had an unstable target knee joint or insufficiently reconstructed ligaments based on medical history and physical examination by the investigator.
* Prohibited medication updated with reference to dosing (formerly screening).

Exclusion Criteria Part A only

* Regular smokers (> 5 cigarettes/day). Urine cotinine levels will be measured during screening for all patients. Regular smokers will be defined as any patient who reports tobacco use of > 5 cigarettes/day and/or who has a urine cotinine ≥ 500 ng/mL.
* Patient had radiologically apparent degenerative joint disease in the target knee as determined by Kellgren and Lawrence grade ≥2 based on X-ray evaluation performed within 9 months from screening.
* Patient had patellofemoral dysplasia Dejour Grade B-D based on X-ray evaluation performed within 9 months from screening
* Patient had malalignment (valgus- or varus-deformity) in the target knee ≥ 5° based on X-ray evaluation performed within 9 months from screening. In suspected cases, the mechanical axis must be established radiographically through complete leg imaging during standing and in postero-anterior (PA) projection.

Exclusion Criteria Part B only

* Regular smokers (> 10 cigarettes/day).
* Clinical signs of inflammation (i.e., redness) in the target knee.
* History of knee replacement (unilateral or total) in either knee.
* Presence of severe hip OA conditioning lower limb function according to PI's evaluation.
* Nephrotic syndrome and/or significant proteinuria
* History of coagulopathy or medical condition requiring anticoagulation which would preclude knee injection
* Patient had malalignment (valgus- or varus-deformity) in the target knee ≥ 7.5° based on X-ray evaluation. In suspected cases, the mechanical axis must be established radiographically through complete leg imaging during standing and in postero-anterior (PA) projection.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2017-09-12 (Actual); Primary Completion 2022-09-06 (Actual); Study Completion 2022-09-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (19):
- United States (11):
  - Novartis Investigative Site, Phoenix, Arizona
  - Novartis Investigative Site, La Mesa, California
  - Novartis Investigative Site, Sacramento, California
  - Novartis Investigative Site, Miami Lakes, Florida
  - Novartis Investigative Site, Sunrise, Florida
  - Novartis Investigative Site, Tampa, Florida
  - Novartis Investigative Site, Boise, Idaho
  - Novartis Investigative Site, Chicago, Illinois
  - Novartis Investigative Site, St Louis, Missouri
  - Novartis Investigative Site, Las Vegas, Nevada
  - Novartis Investigative Site, Philadelphia, Pennsylvania
- Czechia (6):
  - Novartis Investigative Site, Brno, Czech Republic
  - Novartis Investigative Site, Mladá Boleslav, Czech Republic
  - Novartis Investigative Site, Kladno
  - Novartis Investigative Site, Kolín
  - Novartis Investigative Site, Pardubice
  - Novartis Investigative Site, Prague
- Denmark (2):
  - Novartis Investigative Site, Aarhus C
  - Novartis Investigative Site, Hvidovre

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- See also: A Plain Language Trial Summary is available on novctrd.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=2085

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 142 participants were randomized, but only 141 received treatment. One participant in Part B was discontinued due to poor veins that were not adequate for blood samples.
Groups:
- LNA043 20 mg Part A: Part A: a single intra-articular injection of 20 mg LNA043 was administered weekly for 4 weeks for participants with focal cartilage lesions of the knee.
- Placebo Part A: Part A: a single intra-articular injection of matching placebo (0 mg) was administered weekly for 4 weeks for participants with focal cartilage lesions of the knee
- LNA043 20 mg Part B: Part B: a single intra-articular injection of 20 mg LNA043 was administered every 4 weeks from Week 1 to Week 13 (4 injections) for participants with osteoarthritis.
- LNA043 40 mg Part B: Part B: a single intra-articular injection of 40 mg LNA043 was administered every 4 weeks from Week 1 to Week 13 (4 injections) for participants with osteoarthritis.
- Placebo Part B: Part B: a single intra-articular injection of matching placebo (0 mg) was administered every 4 weeks from Week 1 to Week 13 (4 injections) for participants with osteoarthritis
Period: Treatment Period Part A and Part B
Arm/Group | LNA043 20 mg Part A | Placebo Part A | LNA043 20 mg Part B | LNA043 40 mg Part B | Placebo Part B
Started | 43 | 15 | 27 | 27 | 29
Completed | 42 | 15 | 27 | 26 | 29
Not Completed | 1 | 0 | 0 | 1 | 0
Not completed — PI decision based on poor veins for blood sampling | 0 | 0 | 0 | 1 | 0
Not completed — Patient discontinued treatment and entered follow-up | 1 | 0 | 0 | 0 | 0
Period: Post-treatment Follow-up Parts A and B
Arm/Group | LNA043 20 mg Part A | Placebo Part A | LNA043 20 mg Part B | LNA043 40 mg Part B | Placebo Part B
Started | 41 | 15 | 27 | 26 | 29
Completed | 39 | 15 | 24 | 25 | 28
Not Completed | 2 | 0 | 3 | 1 | 1
Not completed — Lost to Follow-up | 1 | 0 | 2 | 0 | 1
Not completed — No longer required treatment | 0 | 0 | 0 | 1 | 0
Not completed — Subject/guardian decision | 1 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | LNA043 20 mg Part A | Placebo Part A | LNA043 20 mg Part B | LNA043 40 mg Part B | Placebo Part B | Total
Number analyzed (Participants) | 43 | 15 | 27 | 27 | 29 | 141
Age, Customized [Number; unit: participants] — Population: Category breakdown for age differed for Part A and Part B
  participants
    ≥18 and ≤55 years Part A only: number analyzed (Participants) | 43 | 15 | 0 | 0 | 0 | 58
    ≥18 and ≤55 years Part A only | 43 | 15 |  |  |  | 58
    ≥18 and ≤64 Part B only: number analyzed (Participants) | 0 | 0 | 27 | 27 | 29 | 83
    ≥18 and ≤64 Part B only |  |  | 18 | 15 | 15 | 48
    ≥65 and ≤76 years - Part B only: number analyzed (Participants) | 0 | 0 | 27 | 27 | 29 | 83
    ≥65 and ≤76 years - Part B only |  |  | 9 | 12 | 14 | 35
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 5 | 19 | 20 | 21 | 86
  Male | 22 | 10 | 8 | 7 | 8 | 55
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 1 | 1 | 0 | 0 | 1 | 3
  White | 42 | 11 | 20 | 26 | 24 | 123
  American Indian or Alaska Native | 0 | 1 | 0 | 0 | 0 | 1
  Black or African | 0 | 1 | 7 | 1 | 3 | 12
  American Unknow | 0 | 1 | 0 | 0 | 0 | 1
  Other | 0 | 0 | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Articular Cartilage Collagen Organization in the Overall Cartilage (Femoral and Patellar Lesions) - Part A
Description: Collagen fibril organization in articular cartilage evaluated by Magnetic Resonance Imaging (MRI) from the cartilage mean T2 relaxation time (with lower values indicative of higher quality). The area of interest is the focal cartilage lesion.
Time Frame: Baseline up to Week 16, Week 28
Population: Pharmacodynamic (PD) analysis set: Subjects with available PD data
Measure: Mean (Standard Error); unit: ms
Arm/Group | LNA043 20 mg Part A | Placebo Part A
Number analyzed (Participants) | 43 | 15
ms
  Week 16 n=43,14: number analyzed (Participants) | 43 | 14
  Week 16 n=43,14 | 3.28 (9.78) | 2.79 (16.37)
  Week 28 n=39,15: number analyzed (Participants) | 39 | 15
  Week 28 n=39,15 | 5.66 (9.90) | 1.98 (15.97)
Statistical Analysis 1: Comparison: LNA043 20 mg Part A vs Placebo Part A; Week 16; Test type: Superiority; Mixed Models Analysis; Mean Difference (Net) = 0.48, 90% CI 2-sided [-30.73 to 31.69]
Statistical Analysis 2: Comparison: LNA043 20 mg Part A vs Placebo Part A; Week 28; Test type: Superiority; Mixed Models Analysis; Mean Difference (Net) = 3.68, 90% CI 2-sided [-27.04 to 34.40]

2. Primary Outcome: Change From Baseline in Articular Cartilage Collagen Organization in the Deep Cartilage Layer (Femoral and Patellar Lesions) - Part A
Description: Collagen fibril organization in articular cartilage evaluated by MRI from the cartilage mean T2 relaxation time (with lower values indicative of higher quality). The area of interest is the focal cartilage lesion.
Time Frame: Baseline up to Week 16, Week 28
Population: Pharmacodynamic (PD) analysis set: Subjects with available PD data
Measure: Mean (Standard Error); unit: ms
Arm/Group | LNA043 20 mg Part A | Placebo Part A
Number analyzed (Participants) | 41 | 15
ms
  Week 16 n=41,14: number analyzed (Participants) | 41 | 14
  Week 16 n=41,14 | 5.30 (9.17) | 3.61 (15.46)
  Week 28 n=39,15: number analyzed (Participants) | 39 | 15
  Week 28 n=39,15 | 7.86 (9.36) | 1.90 (15.08)
Statistical Analysis 1: Comparison: LNA043 20 mg Part A vs Placebo Part A; Week 16; Test type: Superiority; Mixed Models Analysis; Mean Difference (Final Values) = 1.69, 90% CI 2-sided [-27.70 to 31.08]
Statistical Analysis 2: Comparison: LNA043 20 mg Part A vs Placebo Part A; Week 28; Test type: Superiority; Mixed Models Analysis; Mean Difference (Net) = 5.97, 90% CI 2-sided [-23.03 to 34.97]

3. Primary Outcome: Change From Baseline in Articular Cartilage Collagen Organization in the Superficial Cartilage Layer (Femoral and Patellar Lesions) - Part A
Description: Collagen fibril organization in articular cartilage evaluated by MRI from the cartilage mean T2 relaxation time (with lower values indicative of higher quality).The area of interest is the focal cartilage lesion.
Time Frame: Baseline up to Week 16, Week 28
Population: Pharmacodynamic (PD) analysis set: Subjects with available PD data
Measure: Mean (Standard Error); unit: ms
Arm/Group | LNA043 20 mg Part A | Placebo Part A
Number analyzed (Participants) | 17 | 9
ms
  Week 16 n=17,7: number analyzed (Participants) | 17 | 7
  Week 16 n=17,7 | -13.05 (15.68) | -13.93 (24.73)
  Week 28 n=16,9: number analyzed (Participants) | 16 | 9
  Week 28 n=16,9 | -10.45 (16.61) | -12.73 (22.09)
Statistical Analysis 1: Comparison: LNA043 20 mg Part A vs Placebo Part A; Week 16; Test type: Superiority; Mixed Models Analysis; Mean Difference (Net) = 0.88, 90% CI 2-sided [-47.27 to 49.04]
Statistical Analysis 2: Comparison: LNA043 20 mg Part A vs Placebo Part A; Week 28; Test type: Superiority; Mixed Models Analysis; Mean Difference (Net) = 2.27, 90% CI 2-sided [-43.11 to 47.65]

4. Primary Outcome: Change From Baseline of LNA043 to Placebo in Cartilage Volume in the Femoral Medial Index Region (mm3) - Part B
Description: MRI based quantitative assessment using an automated segmentation algorithm
Time Frame: Baseline, Week 29, Week 53
Population: Pharmacodynamic (PD) analysis set: participants with baseline and at least one follow-up MRI assessments for volume of sufficient quality
Measure: Mean (Standard Error); unit: mm^3
Arm/Group | LNA043 20 mg Part B | LNA043 40 mg Part B | Placebo Part B
Number analyzed (Participants) | 12 | 13 | 13
mm^3
  Week 29 n=12,13,13 | 45.52 (61.90) | -12.79 (60.38) | -154.7 (60.25)
  Week 53 n=11,13,7: number analyzed (Participants) | 11 | 13 | 7
  Week 53 n=11,13,7 | 75.64 (54.48) | -36.52 (51.21) | -152.7 (67.72)
Statistical Analysis 1: Comparison: LNA043 20 mg Part B vs Placebo Part B; Test type: Superiority — Week 29; p = 0.0131, Mixed Models Analysis; Mean Difference (Net) = 200.18, 90% CI 2-sided [54.53 to 345.83]
Statistical Analysis 2: Comparison: LNA043 40 mg Part B vs Placebo Part B; Week 29; Test type: Superiority; p = 0.0544, Mixed Models Analysis; Mean Difference (Net) = 141.87, 90% CI 2-sided [-3.83 to 287.56]
Statistical Analysis 3: Comparison: LNA043 20 mg Part B vs Placebo Part B; Week 53; Test type: Superiority; p = 0.0067, Mixed Models Analysis; Mean Difference (Net) = 228.27, 90% CI 2-sided [80.87 to 375.67]
Statistical Analysis 4: Comparison: LNA043 40 mg Part B vs Placebo Part B; Week 53; Test type: Superiority; p = 0.0931, Mixed Models Analysis; Mean Difference (Net) = 116.21, 90% CI 2-sided [-29.52 to 261.94]

5. Primary Outcome: Change From Baseline of LNA043 to Placebo in Cartilage Thickness in the Femoral Medial Index Region (mm) - Part B
Description: MRI based quantitative assessment using an automated segmentation algorithm.
Time Frame: Baseline, Week 29, Week 53
Population: Pharmacodynamic (PD) analysis set: participants with baseline and at least one follow-up MRI assessments for thickness of sufficient quality
Measure: Mean (Standard Error); unit: mm
Arm/Group | LNA043 20 mg Part B | LNA043 40 mg Part B | Placebo Part B
Number analyzed (Participants) | 12 | 13 | 13
mm
  Week 29 n=12,13,13 | 0.01 (0.02) | 0.02 (0.02) | -0.04 (0.02)
  Week 53 n=11,13,7: number analyzed (Participants) | 11 | 13 | 7
  Week 53 n=11,13,7 | -0.01 (0.02) | -0.00 (0.02) | -0.02 (0.03)
Statistical Analysis 1: Comparison: LNA043 20 mg Part B vs Placebo Part B; Week 29; Test type: Superiority; p = 0.0574, Mixed Models Analysis; Mean Difference (Net) = 0.05, 90% CI 2-sided [-0.00 to 0.10]
Statistical Analysis 2: Comparison: LNA043 40 mg Part B vs Placebo Part B; Week 29; Test type: Superiority; p = 0.0248, Mixed Models Analysis; Mean Difference (Net) = 0.06, 90% CI 2-sided [0.01 to 0.11]
Statistical Analysis 3: Comparison: LNA043 20 mg Part B vs Placebo Part B; Week 53; Test type: Superiority; p = 0.3864, Mixed Models Analysis; Mean Difference (Net) = 0.01, 90% CI 2-sided [-0.05 to 0.07]
Statistical Analysis 4: Comparison: LNA043 40 mg Part B vs Placebo Part B; Week 53; Test type: Superiority; p = 0.3290, Mixed Models Analysis; Mean Difference (Net) = 0.02, 90% CI 2-sided [-0.05 to 0.08]

6. Secondary Outcome: Change From Baseline of LNA043 to Placebo in Cartilage Defect Volume (mm^3) for Both Groups of Patients (Femoral and Patellar Lesions) - Part A
Description: Cartilage volume data were generated from the manual segmentation of the cartilage defect that was identified in MR images.
Time Frame: Baseline up to Week 16, Week 28
Population: Pharmacodynamic (PD) analysis set: Subjects with available PD data
Measure: Mean (Standard Error); unit: mm^3
Arm/Group | LNA043 20 mg Part A | Placebo Part A
Number analyzed (Participants) | 40 | 15
mm^3
  Week 16 n=40,14: number analyzed (Participants) | 40 | 14
  Week 16 n=40,14 | -2.42 (8.27) | -7.17 (13.64)
  Week 28 n=39,15: number analyzed (Participants) | 39 | 15
  Week 28 n=39,15 | -11.88 (8.27) | -4.57 (13.45)
Statistical Analysis 1: Comparison: LNA043 20 mg Part A vs Placebo Part A; Week 16; Test type: Superiority; p = 0.6184, Mixed Models Analysis; Mean Difference (Net) = 4.75, 90% CI 2-sided [-21.36 to 30.85]
Statistical Analysis 2: Comparison: LNA043 20 mg Part A vs Placebo Part A; Week 28; Test type: Other; p = 0.3194, Mixed Models Analysis; Mean Difference (Net) = -7.32, 90% CI 2-sided [-33.16 to 18.53]

7. Secondary Outcome: Change From Baseline in Cartilage Mean T2 Relaxation Time as a Marker of Collagen Organization in the Medial Femoral Index Region - Overall Part B
Description: Collagen fibril organisation in articular cartilage evaluated by MRI from the cartilage mean T2 relaxation time (with lower values indicative of higher quality). The area of interest is the femoral medial index region comprising the anterior, central and posterior aspects of the femoral condyle.
Time Frame: Baseline, Week 29, Week 53
Population: Pharmacodynamic (PD) analysis set: Subjects with available PD data
Measure: Mean (Standard Error); unit: ms
Arm/Group | LNA043 20 mg Part B | LNA043 40 mg Part B | Placebo Part B
Number analyzed (Participants) | 27 | 27 | 29
ms
  Week 29 n=21,21,25: number analyzed (Participants) | 21 | 21 | 25
  Week 29 n=21,21,25 | -1.59 (2.25) | -5.07 (2.26) | -4.97 (2.07)
  Week 53 n=20,22,22: number analyzed (Participants) | 20 | 22 | 22
  Week 53 n=20,22,22 | -4.23 (2.29) | -10.53 (2.25) | -3.09 (2.18)
Statistical Analysis 1: Comparison: LNA043 20 mg Part B vs Placebo Part B; Week 29; Test type: Superiority; Mixed Models Analysis; Mean Difference (Net) = 3.38, 90% CI 2-sided [-1.72 to 8.47]
Statistical Analysis 2: Comparison: LNA043 40 mg Part B vs Placebo Part B; Week 29; Test type: Superiority; Mixed Models Analysis; Mean Difference (Net) = -0.10, 90% CI 2-sided [-5.22 to 5.01]
Statistical Analysis 3: Comparison: LNA043 20 mg Part B vs Placebo Part B; Week 53; Test type: Superiority; Mixed Models Analysis; Mean Difference (Net) = -1.14, 90% CI 2-sided [-6.42 to 4.15]
Statistical Analysis 4: Comparison: LNA043 40 mg Part B vs Placebo Part B; Week 53; Test type: Superiority; Mixed Models Analysis; Mean Difference (Net) = -7.44, 90% CI 2-sided [-12.68 to -2.20]

8. Secondary Outcome: Change From Baseline in Cartilage Mean T2 Relaxation Time as a Marker of Collagen Organization in the Medial Femoral Index Region - Deep Part B
Description: as for outcome 7
Time Frame: Baseline, Week 29, Week 53
Population: Pharmacodynamic (PD) analysis set: Subjects with available PD data
Measure: Mean (Standard Error); unit: ms
Arm/Group | LNA043 20 mg Part B | LNA043 40 mg Part B | Placebo Part B
Number analyzed (Participants) | 27 | 27 | 29
ms
  Week 29 n=21,21,25: number analyzed (Participants) | 21 | 21 | 25
  Week 29 n=21,21,25 | -3.80 (2.47) | -5.07 (2.49) | -5.89 (2.26)
  Week 53 n=20,22,22: number analyzed (Participants) | 20 | 22 | 22
  Week 53 n=20,22,22 | -3.93 (2.53) | -12.17 (2.54) | -6.21 (2.41)
Statistical Analysis 1: Comparison: LNA043 20 mg Part B vs Placebo Part B; Week 29; Test type: Superiority; Mixed Models Analysis; Mean Difference (Net) = 2.09, 90% CI 2-sided [-3.49 to 7.66]
Statistical Analysis 2: Comparison: LNA043 40 mg Part B vs Placebo Part B; Week 29; Test type: Superiority; Mixed Models Analysis; Mean Difference (Net) = 0.82, 90% CI 2-sided [-4.82 to 6.45]
Statistical Analysis 3: Comparison: LNA043 20 mg Part B vs Placebo Part B; Week 53; Test type: Superiority; Mixed Models Analysis; Mean Difference (Net) = 2.29, 90% CI 2-sided [-3.54 to 8.11]
Statistical Analysis 4: Comparison: LNA043 40 mg Part B vs Placebo Part B; Week 53; Test type: Superiority; Mixed Models Analysis; Mean Difference (Net) = -5.96, 90% CI 2-sided [-11.81 to -0.10]

9. Secondary Outcome: Change From Baseline in Cartilage Mean T2 Relaxation Time as a Marker of Collagen Organization in the Medial Femoral Index Region - Superficial Part B
Description: as for outcome 7
Time Frame: Baseline, Week 29, Week 53
Population: Pharmacodynamic (PD) analysis set: Subjects with available PD data
Measure: Mean (Standard Error); unit: ms
Arm/Group | LNA043 20 mg Part B | LNA043 40 mg Part B | Placebo Part B
Number analyzed (Participants) | 27 | 27 | 29
ms
  Week 29 n=21,21,25: number analyzed (Participants) | 21 | 21 | 25
  Week 29 n=21,21,25 | -0.06 (2.51) | -4.16 (2.51) | -3.53 (2.30)
  Week 53 n=20,22,22: number analyzed (Participants) | 20 | 22 | 22
  Week 53 n=20,22,22 | -3.54 (2.36) | -9.07 (2.36) | -0.91 (2.25)
Statistical Analysis 1: Comparison: LNA043 20 mg Part B vs Placebo Part B; Week 29; Test type: Superiority; Mixed Models Analysis; Mean Difference (Net) = 3.47, 90% CI 2-sided [-2.21 to 9.15]
Statistical Analysis 2: Comparison: LNA043 40 mg Part B vs Placebo Part B; Week 29; Test type: Superiority; Mixed Models Analysis; Mean Difference (Net) = -0.63, 90% CI 2-sided [-6.31 to 5.04]
Statistical Analysis 3: Comparison: LNA043 20 mg Part B vs Placebo Part B; Week 53; Test type: Superiority; Mixed Models Analysis; Mean Difference (Net) = -2.63, 90% CI 2-sided [-8.07 to 2.82]
Statistical Analysis 4: Comparison: LNA043 40 mg Part B vs Placebo Part B; Week 53; Test type: Superiority; Mixed Models Analysis; Mean Difference (Net) = -8.16, 90% CI 2-sided [-13.61 to -2.72]

10. Secondary Outcome: Incidence of Immunogenicity (IG) Part A
Description: A validated ligand binding assay were used for the detection of anti-LNA043 antibodies, and cross-reactivity to ANGPTL3 and ANGPTL4.
Time Frame: Week 1,3,8,16,28
Population: Safety analysis set
Measure: Number; unit: participants
Arm/Group | LNA043 20 mg Part A | Placebo Part A
Number analyzed (Participants) | 43 | 15
participants
  Week 1 (Day 1) Predose | 0 | 0
  Week 3 (Day 15) Pre-dose | 0 | 0
  Week 8 (Day 50) | 0 | 0
  Week 16 (Day 106) | 0 | 0
  Week 28 (Day 190) | 0 | 0

11. Secondary Outcome: Incidence of Immunogenicity (IG) Part B
Description: as for outcome 10
Time Frame: Week 1,5,9,13,17,29,53
Population: Safety analysis set
Measure: Number; unit: participants
Arm/Group | LNA043 20 mg Part B | LNA043 40 mg Part B | Placebo Part B
Number analyzed (Participants) | 27 | 27 | 29
participants
  Week 1 (Day 1) Predose | 0 | 0 | 0
  Week 5 Pre-dose | 0 | 0 | 0
  Week 9 | 0 | 0 | 0
  Week 13 | 0 | 0 | 0
  Week 17 | 0 | 0 | 0
  Week 29 | 0 | 0 | 0
  Week 53 | 0 | 0 | 0

12. Secondary Outcome: Serum Concentrations of LNA043 - Part A
Description: Concentrations for LNA043 were determined by a validated LC-MS/MS method; the anticipated LLOQ was 10ng/mL in serum. Concentrations below the LLOQ were reported as "zero"
Time Frame: Week 1: 0 (pre-dose), 0.25 hours, 1, 2 hours post dose; Weeks 2, 3, 4: 0 hour (pre dose), 1 hour post dose
Population: Pharmacokinetic analysis set
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | LNA043 20 mg Part A
Number analyzed (Participants) | 43
ng/mL
  Week 1, 0 hour pre-dose | 0 (0)
  Week 1, 0.25 hour post dose n=6: number analyzed (Participants) | 6
  Week 1, 0.25 hour post dose n=6 | 24.9 (16.3)
  Week 1, 1 hour post dose n=7: number analyzed (Participants) | 7
  Week 1, 1 hour post dose n=7 | 65.1 (30.2)
  Week 1, 2 hours post dose n=41: number analyzed (Participants) | 41
  Week 1, 2 hours post dose n=41 | 64.9 (37.5)
  Week 2,0 hour pre dose n=42: number analyzed (Participants) | 42
  Week 2,0 hour pre dose n=42 | 0.00 (0.00)
  Week 2, 1 hour post dose n=43 | 48.1 (32.9)
  Week 3, 0 hour pre dose n=41: number analyzed (Participants) | 41
  Week 3, 0 hour pre dose n=41 | 0.00 (0.00)
  Week 3, 1 hour post dose n=39: number analyzed (Participants) | 39
  Week 3, 1 hour post dose n=39 | 51.0 (37.6)
  Week 4, 0 hour pre dose n=42: number analyzed (Participants) | 42
  Week 4, 0 hour pre dose n=42 | 3.00 (19.4)
  Week 4, 1 hour post dose n=41: number analyzed (Participants) | 41
  Week 4, 1 hour post dose n=41 | 52.9 (38.1)

13. Secondary Outcome: Serum Concentrations of ANGPTL3 - Part A
Description: Validated bioanalytical assays were used to determine ANGPTL3 in serum with an LLOQ of 2.13 ng/mL. Concentrations below the LLOQ were reported as "zero"
Time Frame: Week 1: 0 (pre-dose), 0.25 hours, 1, 2 hours post dose; Weeks 2, 3, 4: 0 hour (pre dose), 1 hour post dose
Population: Pharmacokinetic analysis set
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | LNA043 20 mg Part A | Placebo Part A
Number analyzed (Participants) | 43 | 15
ng/mL
  Week 1, 0 hour pre-dose n=41,14: number analyzed (Participants) | 41 | 14
  Week 1, 0 hour pre-dose n=41,14 | 19.1 (9.29) | 23.3 (8.55)
  Week 1, 0.25 hour post dose n=6,2: number analyzed (Participants) | 6 | 2
  Week 1, 0.25 hour post dose n=6,2 | 20.8 (8.12) | 20.4 (6.36)
  Week 1, 1 hour post dose n=7,2: number analyzed (Participants) | 7 | 2
  Week 1, 1 hour post dose n=7,2 | 19.7 (8.65) | 18.2 (3.32)
  Week 1, 2 hours post dose n=40,15: number analyzed (Participants) | 40 | 15
  Week 1, 2 hours post dose n=40,15 | 18.9 (9.38) | 24.3 (9.52)
  Week 2,0 hour pre dose n=42,15: number analyzed (Participants) | 42 | 15
  Week 2,0 hour pre dose n=42,15 | 18.9 (10.3) | 21.7 (10.2)
  Week 2, 1 hour post dose n=42,15: number analyzed (Participants) | 42 | 15
  Week 2, 1 hour post dose n=42,15 | 18.3 (8.06) | 19.7 (9.58)
  Week 3, 0 hour pre dose n=42,14: number analyzed (Participants) | 42 | 14
  Week 3, 0 hour pre dose n=42,14 | 19.1 (7.79) | 24.2 (9.95)
  Week 3, 1 hour post dose n=39,14: number analyzed (Participants) | 39 | 14
  Week 3, 1 hour post dose n=39,14 | 18.5 (7.35) | 28.9 (16.4)
  Week 4, 0 hour pre dose n=42,15: number analyzed (Participants) | 42 | 15
  Week 4, 0 hour pre dose n=42,15 | 19.6 (8.71) | 21.0 (7.11)
  Week 4, 1 hour post dose n=41,15: number analyzed (Participants) | 41 | 15
  Week 4, 1 hour post dose n=41,15 | 19.6 (7.87) | 22.6 (9.06)

14. Secondary Outcome: Synovial Fluid Concentrations of LNA043 - Part A
Description: Concentrations for LNA043 were determined by a validated LC-MS/MS method; the anticipated LLOQ was 10ng/mL in synovial fluid. Concentrations below the LLOQ were reported as "zero".
Time Frame: Weeks 1,2,3,4: 0 hour (pre-dose)
Population: LNA043 Stability in synovial fluid could not be demonstrated. Consequently, the assay was not considered suitable for the determination of LNA043 in synovial fluid collected in Part A and no reportable concentrations of LNA043 in synovial fluid are available in Part A, samples were never assayed and so data are not available for LNA043 concentrations in synovial fluid for Part A.
Arm/Group | LNA043 20 mg Part A
Number analyzed (Participants) | 0

15. Secondary Outcome: Synovial Fluid Concentrations of ANGPTL3 - Part A
Description: Validated bioanalytical assays were used to determine ANGPTL3 in synovial fluid with an LLOQ of 2.74 ng/mL. Concentrations below the LLOQ were reported as "zero".
Time Frame: Weeks 1,2,3,4: 0 hour (pre-dose)
Population: Pharmacokinetic analysis set
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | LNA043 20 mg Part A | Placebo Part A
Number analyzed (Participants) | 43 | 15
ng/mL
  Week 1, 0 hour pre-dose n=8,3: number analyzed (Participants) | 8 | 3
  Week 1, 0 hour pre-dose n=8,3 | 0.00 (0.00) | 00.0 (00.0)
  Week 2,0 hour pre dose n=11,5: number analyzed (Participants) | 11 | 5
  Week 2,0 hour pre dose n=11,5 | 0.00 (0.00) | 00.0 (00.0)
  Week 3, 0 hour pre dose n=13,4: number analyzed (Participants) | 13 | 4
  Week 3, 0 hour pre dose n=13,4 | 0.616 (2.22) | 00.0 (00.0)
  Week 4, 0 hour pre dose n=15,3: number analyzed (Participants) | 15 | 3
  Week 4, 0 hour pre dose n=15,3 | 1.42 (5.50) | 00.0 (00.0)

16. Secondary Outcome: Serum Concentrations of LNA043 - Part B
Description: Concentrations for LNA043 were determined by a validated LC-MS/MS method; the anticipated LLOQ was 10ng/mL in serum. Concentrations below the LLOQ were reported as "zero
Time Frame: Week 1: 0 (pre-dose), 2 hours post dose; Weeks 5 and 13: 1 hour post dose
Population: Pharmacokinetic analysis set
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | LNA043 20 mg Part B | LNA043 40 mg Part B
Number analyzed (Participants) | 27 | 27
ng/mL
  Week 1, 0 hours pre-dose n=27,26: number analyzed (Participants) | 27 | 26
  Week 1, 0 hours pre-dose n=27,26 | 3.48 (18.1) | 7.96 (40.6)
  Week 1, 2 hours post dose n=24,24,: number analyzed (Participants) | 24 | 24
  Week 1, 2 hours post dose n=24,24, | 76.4 (51.0) | 158 (94.0)
  Week 5, 1 hour post dose n=27,26: number analyzed (Participants) | 27 | 26
  Week 5, 1 hour post dose n=27,26 | 55.6 (47.0) | 101 (74.2)
  Week 13, 1 hour post dose n=27,25: number analyzed (Participants) | 27 | 25
  Week 13, 1 hour post dose n=27,25 | 59.5 (53.0) | 118 (78.2)

17. Secondary Outcome: Serum Concentrations of ANGPTL3 - Part B
Description: as for outcome 13
Time Frame: Week 1: 0 (pre-dose), 2 hours post dose; Weeks 5 and 13: 1 hour post dose
Population: Pharmacokinetic analysis set
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | LNA043 20 mg Part B | LNA043 40 mg Part B | Placebo Part B
Number analyzed (Participants) | 27 | 26 | 29
ng/mL
  Week 1, 0 hour pre-dose n=27,26,29 | 25.3 (11.1) | 21.9 (9.09) | 26.6 (14.0)
  Week 1, 2 hours post dose n=24,24,26: number analyzed (Participants) | 24 | 24 | 26
  Week 1, 2 hours post dose n=24,24,26 | 26.0 (12.8) | 23.9 (10.6) | 27.6 (13.1)
  Week 5, 1 hour post dose n=26,26,28: number analyzed (Participants) | 26 | 26 | 28
  Week 5, 1 hour post dose n=26,26,28 | 21.8 (9.80) | 23.3 (9.97) | 26.2 (10.8)
  Week 13, 1 hour post dose n=27,25,28: number analyzed (Participants) | 27 | 25 | 28
  Week 13, 1 hour post dose n=27,25,28 | 22.9 (8.72) | 22.5 (8.39) | 24.8 (11.8)

18. Secondary Outcome: Synovial Fluid Concentrations of LNA043 Part B
Description: as for outcome 14
Time Frame: Weeks 1,5.9.13: 0 hour (pre-dose)
Population: Pharmacokinetic analysis set
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | LNA043 20 mg Part B | LNA043 40 mg Part B
Number analyzed (Participants) | 11 | 6
ng/mL
  Week 1, 0 hours pre dose n=9,5: number analyzed (Participants) | 9 | 5
  Week 1, 0 hours pre dose n=9,5 | 28.9 (86.7) | 0.00 (0.00)
  Week 5, 0 hours pre dose n=10,5: number analyzed (Participants) | 10 | 5
  Week 5, 0 hours pre dose n=10,5 | 368 (1160) | 18.1 (40.6)
  Week 9, 0 hours pre-dose n=11,6 | 0.00 (0.00) | 43600 (90900)
  Week 13, 0 hours pre dose n=8,4: number analyzed (Participants) | 8 | 4
  Week 13, 0 hours pre dose n=8,4 | 0.00 (0.00) | 199000 (398000)

19. Secondary Outcome: Synovial Fluid Concentrations of ANGPTL3 - Part B
Description: as for outcome 15
Time Frame: Weeks 1,5.9.13: 0 hour (pre-dose)
Population: Pharmacokinetic analysis set
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | LNA043 20 mg Part B | LNA043 40 mg Part B | Placebo Part B
Number analyzed (Participants) | 10 | 5 | 12
ng/mL
  Week 1, 0 hour pre-dose n=8,3,8: number analyzed (Participants) | 8 | 3 | 8
  Week 1, 0 hour pre-dose n=8,3,8 | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00)
  0.00Week 5,,0 hour pre dose n=10,5,12 | 1.00 (3.16) | 4.38 (9.79) | 1.57 (5.43)
  Week 9,, 0 hour pre dose n=8,4,9: number analyzed (Participants) | 8 | 4 | 9
  Week 9,, 0 hour pre dose n=8,4,9 | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00)
  Week 13, 0 hour pre dose n=7,4,8: number analyzed (Participants) | 7 | 4 | 8
  Week 13, 0 hour pre dose n=7,4,8 | 0.00 (0.00) | 1.87 (3.74) | 0.890 (2.52)

20. Primary Outcome: Overview of Number of Participants With Adverse Events and Serious Adverse Events for Part A and Part B
Description: Treatment emergent other and serious adverse events (TEAE and TESAE) period:
  Part A: Baseline up to Day 50 (included 30 day safety follow-up Part B: Baseline up to Day 113 (included 30 day safety follow-up)
  Long term Follow-UP period:
  Part A: Day 51 to Day 365 Part B: Day 114 to Day 365
Time Frame: Baseline up to end of post treatment follow-up
Population: Safety analysis set
Measure: Number; unit: participants
Groups:
- LNA043 40mg Part B: Part B: a single intra-articular injection of 40 mg LNA043 was administered every 4 weeks from Week 1 to Week 13 (4 injections) for participants with osteoarthritis.
Arm/Group | LNA043 20 mg Part A | Placebo Part A | LNA043 20 mg Part B | LNA043 40mg Part B | Placebo Part B
Number analyzed (Participants) | 43 | 15 | 27 | 27 | 29
participants
  Part A TEAE: number analyzed (Participants) | 43 | 15 | 0 | 0 | 0
  Part A TEAE | 19 | 7 |  |  |
  Part A TESAE: number analyzed (Participants) | 43 | 15 | 0 | 0 | 0
  Part A TESAE | 0 | 0 |  |  |
  Part A - Follow-up AE: number analyzed (Participants) | 41 | 15 | 0 | 0 | 0
  Part A - Follow-up AE | 16 | 1 |  |  |
  Part A - Follow-up SAE: number analyzed (Participants) | 41 | 15 | 0 | 0 | 0
  Part A - Follow-up SAE | 2 | 0 |  |  |
  Part B - TEAE: number analyzed (Participants) | 0 | 0 | 27 | 27 | 29
  Part B - TEAE |  |  | 6 | 15 | 10
  Part B - TESAE: number analyzed (Participants) | 0 | 0 | 27 | 27 | 29
  Part B - TESAE |  |  | 1 | 0 | 0
  Part B - Follow-up AE: number analyzed (Participants) | 0 | 0 | 27 | 26 | 29
  Part B - Follow-up AE |  |  | 1 | 1 | 7
  Part B B - Follow-up SAE: number analyzed (Participants) | 0 | 0 | 27 | 26 | 29
  Part B B - Follow-up SAE |  |  | 1 | 0 | 2

ADVERSE EVENTS:
Time Frame: Treatment emergent (TE) averse events: Part A: Baseline up to Day 50 (including 30 day safety follow-up post last dose) Part B: Baseline up to Day 113 (including 30 day safety follow-up post last dose) Long term Follow-Up (FU) period: Part A: Day 51 to Day 365 Part B: Day 114 to Day 365
Groups:
- LNA043 20 mg Part A - TE: Part A: a single intra-articular injection of 20 mg LNA043 was administered weekly for 4 weeks for participants with focal cartilage lesions of the knee.
  Treatment Emergent (TE) AEs are reported Baseline up to Day 50.
- Placebo Part A - TE: Part A: a single intra-articular injection of matching placebo (0 mg) was administered weekly for 4 weeks for participants with focal cartilage lesions of the knee.
  Treatment Emergent (TE) AEs are reported Baseline up to Day 50.
- LNA043 20 mg Part B - TE: Part B: a single intra-articular injection of 20 mg LNA043 was administered every 4 weeks from Week 1 to Week 13 (4 injections) for participants with osteoarthritis.
  Treatment Emergent (TE) AEs are reported Baseline up to Day 113.
- LNA043 40 mg Part B - TE: Part B: a single intra-articular injection of 40 mg LNA043 was administered every 4 weeks from Week 1 to Week 13 (4 injections) for participants with osteoarthritis.
  Treatment Emergent (TE) AEs are reported Baseline up to Day 113.
- Placebo Part B - TE: Part B: a single intra-articular injection of matching placebo (0 mg) was administered every 4 weeks from Week 1 to Week 13 (4 injections) for participants with osteoarthritis.
  Treatment Emergent (TE) AEs are reported Baseline up to Day 113.
- LNA043 20 mg Part A - FU: Part A: a single intra-articular injection of 20 mg LNA043 was administered weekly for 4 weeks for participants with focal cartilage lesions of the knee.
  AEs in long term Follow-Up (FU) period are reported form Day 51 to Day 365.
- Placebo Part A - FU: Part A: a single intra-articular injection of matching placebo (0 mg) was administered weekly for 4 weeks for participants with focal cartilage lesions of the knee.
  AEs in long term Follow-Up (FU) period are reported form Day 51 to Day 365.
- LNA043 20 mg Part B - FU: Part B: a single intra-articular injection of 20 mg LNA043 was administered every 4 weeks from Week 1 to Week 13 (4 injections) for participants with osteoarthritis.
  AEs in long term Follow-Up (FU) period are reported form Day 114 to Day 365.
- LNA043 40 mg Part B - FU: Part B: a single intra-articular injection of 40 mg LNA043 was administered every 4 weeks from Week 1 to Week 13 (4 injections) for participants with osteoarthritis.
  AEs in long term Follow-Up (FU) period are reported form Day 114 to Day 365.
- Placebo Part B - FU: Part B: a single intra-articular injection of matching placebo (0 mg) was administered every 4 weeks from Week 1 to Week 13 (4 injections) for participants with osteoarthritis.
  AEs in long term Follow-Up (FU) period are reported form Day 114 to Day 365.
Arm/Group | LNA043 20 mg Part A - TE | Placebo Part A - TE | LNA043 20 mg Part B - TE | LNA043 40 mg Part B - TE | Placebo Part B - TE | LNA043 20 mg Part A - FU | Placebo Part A - FU | LNA043 20 mg Part B - FU | LNA043 40 mg Part B - FU | Placebo Part B - FU
All-Cause Mortality (participants affected / at risk) | 0/43 | 0/15 | 0/27 | 0/27 | 0/29 | 0/43 | 0/15 | 0/27 | 0/27 | 0/29
Serious Adverse Events (participants affected / at risk) | 0/43 | 0/15 | 1/27 | 0/27 | 0/29 | 2/43 | 0/15 | 1/27 | 0/27 | 2/29
Other Adverse Events (participants affected / at risk) | 19/43 | 7/15 | 6/27 | 15/27 | 10/29 | 16/43 | 1/15 | 3/27 | 5/27 | 12/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LNA043 20 mg Part A - TE (N=43) | Placebo Part A - TE (N=15) | LNA043 20 mg Part B - TE (N=27) | LNA043 40 mg Part B - TE (N=27) | Placebo Part B - TE (N=29) | LNA043 20 mg Part A - FU (N=43) | Placebo Part A - FU (N=15) | LNA043 20 mg Part B - FU (N=27) | LNA043 40 mg Part B - FU (N=27) | Placebo Part B - FU (N=29)
Blood loss anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Odontogenic cyst (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Colitis ischaemic (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
COVID-19 pneumonia (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vena cava thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LNA043 20 mg Part A - TE (N=43) | Placebo Part A - TE (N=15) | LNA043 20 mg Part B - TE (N=27) | LNA043 40 mg Part B - TE (N=27) | Placebo Part B - TE (N=29) | LNA043 20 mg Part A - FU (N=43) | Placebo Part A - FU (N=15) | LNA043 20 mg Part B - FU (N=27) | LNA043 40 mg Part B - FU (N=27) | Placebo Part B - FU (N=29)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Anaemia macrocytic (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Coronary artery disease (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Homocystinaemia (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Odontogenic cyst (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Thyroid mass (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cataract (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dental caries (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Faecaloma (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gastritis haemorrhagic (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Hiatus hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Large intestine polyp (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Oesophagitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Inflammation (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Injection site bruising (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Injection site erythema (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Injection site haematoma (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Injection site joint erythema (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Injection site joint pain (General disorders) | 2 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Peripheral swelling (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vessel puncture site haemorrhage (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
COVID-19 (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
COVID-19 pneumonia (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gingivitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Herpes zoster (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Infected dermal cyst (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Respiratory tract infection viral (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tonsillitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 2 | 1 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Bone contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Epicondylitis (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Limb injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Meniscus cyst (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Muscle strain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Nail injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Tendon injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tooth fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Traumatic haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 2
Blood pressure increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Blood uric acid increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Cardiac murmur (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Haematology test abnormal (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hepatic enzyme increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
SARS-CoV-2 test positive (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Urine protein/creatinine ratio increased (Investigations) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 1 | 1 | 4 | 1 | 3 | 0 | 0 | 2 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Chondropathy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 4 | 0 | 1 | 1 | 3 | 0 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Osteopenia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 6 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Seizure (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Sleep disorder (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Microalbuminuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Atrophic vulvovaginitis (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Breast pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Ovulation pain (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Lichenoid keratosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Haematoma (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Varicose vein (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0

LIMITATIONS AND CAVEATS:
For several outcomes there was a loss in samples size, which may limit the interpretability of results. For Part B, subgroup 1 was defined to address heterogeneity in MRI quality, and to ensure validity of the reported data. P-values for T2 relaxation time are omitted, as there was an error in the calculation. For Part A, the protocol sample size section refers to a ratio for the primary analysis, but data was reported as superficial and deep cartilage layers separately. Both will be updated.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2020-12-22): https://cdn.clinicaltrials.gov/large-docs/64/NCT03275064/Prot_000.pdf
  • Statistical Analysis Plan (2022-12-05): https://cdn.clinicaltrials.gov/large-docs/64/NCT03275064/SAP_001.pdf